CLINICAL TRIAL: NCT03757793
Title: Near-infrared Spectroscopy for Monitoring Tissue Oxygenation in Breast Reconstruction
Status: Terminated | Type: Observational
Why Stopped: It is practically not feasible to maintain the electrodes in place for 72 hours.
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Joke De Wachter, data manager, University Hospital, Antwerp
Other Study IDs: 18/12/173
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mastectomy; Breast Reconstruction; Flap Ischemia
Keywords: Near infrared spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Reliability of NIRS in DIEP flap surgery: In patients who underwent DIEP flap surgery, monitoring of postoperative tissue oxygen saturation of the flap by use of the FORE-SIGHT Elite monitor will be compared to standard of care physical examination.
  Interventions: Device: FORE-SIGHT ELITE monitor

INTERVENTIONS:
Device: FORE-SIGHT ELITE monitor — At end of surgery, one sensor of the FORE-SIGHT Elite monitor is placed on the DIEP flap or two sensors in case of bilateral DIEP flaps for monitoring perfusion and oxygen consumption in the free flap. A control sensor of the FORE-SIGHT Elite monitor placed on the abdomen where tissue is taken to perform the DIEP flap. This sensor reflects normal tissue oxygenation. Data obtained from the FORE-SIGHT Elite monitor will be compared to data obtained from physical examination, which is standard of care for flap monitoring.

SUMMARY:
The study will evaluate the use of near infrared spectrometry (NIRS)in detecting early microvascular complications in deep inferior epigastric artery perforator (DIEP)-flap(s).

DETAILED DESCRIPTION:
After a complex resection for breast cancer (e.g. mastectomy), a microvascular flap reconstruction can be used to fill up the tissue defects. A deep inferior epigastric artery perforator (DIEP)-flap is one of the most used microvascular flap reconstructions. Skin and fat from the abdomen are used to reconstruct a new breast.The success ratio of this type of surgery is high, more than 95%. Nevertheless, free flap failure can have disastrous consequences.The flap can be injured by surgical factors such as vascular complications.This is one of the major concerns and it usually occurs in the first hours after surgery. The success rate of the free flap depends on the continuous arterial inflow and the venous outflow through the new microvascular anastomoses. Thrombosis, kinking or external compression on the micro- and macrovascular blood vessels can cause necrosis of the flap. It is essential to recognize these complications as fast as possible to maximize the potential for flap salvage. Physical examination is still the gold standard for flap monitoring. However this monitoring is subjective, labor intensive and requires experience. Because of these disadvantages, a more objective method is desirable. In this suggested project, the flap will be monitored with FORE-SIGHT ELITE monitor( CAS Medical Systems incorporated) during the first 72 hours postoperatively. In this period most complications occur. The FORE-SIGHT ELITE Absolute Tissue Oximeter is a non-invasive device that measures absolute tissue oxygen saturation. It operates on the principle that blood contains hemoglobin in two primary forms, oxygenated hemoglobin (HbO2 ) and de-oxygenated hemoglobin (Hb), which absorb near-infrared light in different, measurable ways.The FORE-SIGHT ELITE incorporates CAS Medical Systems exclusive technology to project harmless near-infrared light in five precise wavelengths (690, 730, 770, 810 and 870 nanometer). An algorithm analyzes the reflected wavelengths. The algorithm is specially designed for the tissue with attention to unique characteristics of the tissue. Reflected light is captured by detectors positioned on the sensor for optimal signal collection. After analyzing the reflected light, the FORE-SIGHT ELITE displays the tissue oxygen saturation level on the monitor as an absolute number and provides a graphical representation of historical values.The FORE-SIGHT ELITE has been validated to determine cerebral tissue oxygen saturation amongst other in brain surgery. Tissue oxygen saturation (StO2) levels are determined by the ratio of oxygenated hemoglobin to total hemoglobin at the microvascular level (arterioles, venules, and capillaries) in the region to which the sensor is applied. This technique is called Near Infrared Spectroscopy (NIRS).Validated use of NIRS would be a major advantage to detect ischaemia in DIEP flaps. In the study pediatric sensor size is used to ensure proper depth of light penetration in a limited operating zone. By application of small neonatal sensors ( Foresight®-sensors (CASMED, Branford, CT, USA), on unilateral or bilateral DIEP flaps,light penetrates at 1.25cm depth.This reflects the perfusion and the oxygen consumption in the free flap.

A control pediatric sensor is placed on the abdomen where tissue is taken to perform the DIEP flap. This sensor reflects the normal tissue oxygenation of the patient. NIRS uses this technology for the detection of ischemia and hypoxia. It is a real-time, continuous, non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective unilateral or bilateral breast reconstruction via DIEP flap procedure.

Exclusion Criteria:

* refusal of written informed consent
* redo-surgery
* known history of allergy to adhesives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, over 18 years, undergoing unilateral or bilateral DIEP flap procedure
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Detection of ischaemia after DIEP flap surgery by use of NIRS | first 72 hours post surgery
  The aim of the study is to determine whether near infrared spectrometry(NIRS) would be a validated tool to detect early microvascular complications. A decrease of 10% of the Sct O2 taken at the DIEP flap(s) compared to Sct O2 of the abdomen will be considered as possible risk of ischaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium